CLINICAL TRIAL: NCT01455792
Title: MRI and Ultrasound Soft Image Fusion Guided Biopsies Compared to Gold Standard Prostate Biopsies
Brief Title: Biopsy Study Comparing MRI and Ultrasound Soft Image Fusion Guided Biopsies and Gold Standard Prostate Biopsies.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Erik Rud, Attending radiologist, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-09143c2009/2183
Record Dates: First submitted 2011-09-20; First posted 2011-10-20 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer
Keywords: Biopsy; MRI and ultrasound soft image fusion; Gold standard TRUS biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI and soft image fusion biopsy (Experimental): Preoperative MRI and soft image ultrasound guided biopsy.
  Interventions: Procedure: Biopsies using image fusion
- Gold standard biopsy (Active Comparator): Gold standard TRUS biopsy
  Interventions: Procedure: Biopsies using image fusion; Procedure: Gold standard biopsy

INTERVENTIONS:
Procedure: Biopsies using image fusion — MRI and soft image fusion guided biopsy
  Other Names: Urostation,Koelis,Grenoble, France
Procedure: Gold standard biopsy — Gold standard TRUS biopsy
  Other Names: Gold standard
  Arms: Gold standard biopsy

SUMMARY:
Background: Prostate biopsies are usually performed due to accidentally discovered elevated prostate specific antigen (PSA) and/or abnormal digital rectal examination. Transrectal ultrasound (TRUS) guided biopsy is standard procedure, but possibility for precise documentation concerning the localization of the biopsies are lacking. Therefore, the same locations might be subject to multiple negative biopsies. There is a growing confidence that magnetic resonance imaging (MRI) of the prostate gland can identify significant, high-grade tumours, and studies have shown value in performing MRI before biopsies. Because image documentation is lacking, it is not possible to know which region actually being biopsied with conventional TRUS biopsy. MRI and 3D ultrasound soft image fusion guided biopsy, is a new promising method that will ascertain all regions of the prostate gland to be biopsied, and it is possible to perform accurate targeted biopsies when combined with MRI.

Aims of the study

Compare the biopsy results in the two groups:

1. To evaluate the overall rate of positive biopsies.
2. To evaluate the rate of re-biopsies.
3. To evaluate the detection rate of Gleason grade 4 and 5 tumours.
4. To evaluate the rate of positive targeted biopsies.
5. To evaluate the rate of positive random biopsies
6. To compare targeted and random biopsies between groups.
7. To compare patient tolerance, time consumption and cost of the two methods.
8. To evaluate the diagnostic accuracy of performing cytological imprints of targeted biopsies.

Material and methods: A prospective randomized study including 300 consecutive patients referred to the initial biopsy. The patients are randomized to conventional TRUS biopsies and image fusion guided biopsy.

All patients undergo a minimum 12-core re-biopsy procedure. In addition a targeted biopsy will be obtained in case of positive MRI of ultrasound.

DETAILED DESCRIPTION:
Biopsy procedures

1. Conventional TRUS biopsy procedure (Gold standard). These patients will first undergo 0-6 TRUS targeted biopsies (TRUS TB) (2 targeted biopsies in up to 3 lesions), directed towards lesions suspect of prostate cancer seen on TRUS, or detected by DRE (standard-target). Subsequently, they will undergo a standard random 12 core TRUS guided biopsy procedure. All biopsies will be performed using the Bruel and Kjaer ultrasound unit, type 1846, and transrectal transducer No 8531 (New york, United States). If there for any reason would be desirable to reduce the total number of biopsies, we will omit random biopsies if targeted biopsies already have been taken at that specific site.

   Two dedicated urologist, (L. M. E. and G. M.), with special interest and experience in prostate cancer will perform conventional TRUS biopsies according to the protocol, and according to their previous experience. No effort will be done for these two urologists to harmonize their biopsy procedures.
2. 3D image documented biopsy (3D IDB) procedure. These patients will first undergo an MRI examination of the prostate. Possible cancer-suspect areas will be identified and mapped in 3D. MRI findings with high grade of cancer suspicion will be marked as red circles with diameter from 6 to 8 mm. MRI finding compatible with low or intermediate cancer suspicions will be labelled as yellow circles from 6 to 8 mm in the diameter. The circles will be placed in the centre of MRI findings. A few days later the patients will first undergo 0-6 targeted biopsies, directed towards possible lesions detected by MRI, which are transferred (by soft image fusion) to the TRUS images, allowing for TRUS biopsies directed towards lesions detected by MRI, so-called MRI targeted biopsies (MRI TB). These biopsies will be used for additional cytological imprints for evaluation of presence/absence of carcinoma.

Subsequently, they will undergo 12 core random TRUS guided biopsy procedure, using the 3D IDB software and 3D TRUS equipment (3D IDB random). When performing these random biopsies, the MRI findings will not be displayed on the US screen.

One dedicated urologist (E. B.) with substantial experience with the 3D IDB procedure will perform the MRI TB.

Biopsy procedures will be performed in local anaesthesia using 6-10 ml 2% Lidocaine. Using ultrasound control, local anaesthetic is injected around the prostate using a 22-gauge spinal needle. Prostate volume is calculated using the standard ellipsoid formula, multiplying the largest anterioposterior (height), transverse (width) and cephalocaudal (length) prostate diameters by 0,524.

Biopsies will be performed using 18 gauge spring-loaded needle (Angiotech®). All individual biopsies cores will be marked and kept in separate glasses for fixation.

Biopsy time defined as time when the TRUS probe is in place is registered in both groups.

MRI examination Patients randomized to the 3D IDB procedure with MRI US fusion, will undergo examination of the prostate using a 1,5 T MR scanner (Siemens Avanto, Erlangen Germany) with a body array coil. Total scan time will be approximately 12 minutes.

Siemens Picture Archive Communicating System (PACS) and Nordic ICE® will be used for post processing analyses. Evaluation of the MRI examinations will be performed by one radiologist (E. R.).

Patient preparation Warfarin anticoagulant therapy is stopped 3 days before biopsy procedure and biopsy is not performed if international normalized ratio (INR) value is over 2,0. If needed, low molecular weight heparin can be administered to the patient. A cleansing enema is not strictly required. One hour before the biopsy procedure is planned a peroral antibiotic (Trimethoprim 160 mg, Sulfamethoxazole 800 mg) is administered and additional dose is taken the following evening.

Assessment of patient tolerance and discomfort will be registered in both groups by visual analogue score (VAS) pain score questionnaire (10 scores denoting the worst and 0 denoting no bother).

Cytological procedures Each targeted biopsy will be subject to cytological imprint. These smears will undergo standard staining and classified as positive or negative according to presence of carcinoma or not.

Histopathological procedures Routine hematoxylin and eosin (HE) stain of the biopsies will be performed, and evaluated according to Gleason system (gold standard for histological evaluation) ranging from 1-5, with 5 being the most aggressive tumour. Gleason score is the sum of the two dominating Gleason grades, for instance 5+5 for the most aggressive tumour giving a Gleason score of 10. The biopsies will be marked, in order to evaluate the spatial distribution of cancer.

The length of the biopsy core and tumour involvement will be measured.

Null hypotheses

1. There is no difference in the overall prostate cancer detection (rate of positive biopsies) between the group undergoing conventional TRUS biopsy procedure and the group undergoing 3D IDB MRI TB.
2. There is not higher rate of Gleason grade 4 and 5 in the 3D IDB MRI TB group compared to the conventional TRUS group.
3. The 3D IDB MRI TB group do not have more prostate cancer than random 3D IDB
4. The MRI TB does not detect more prostate cancer than TRUS TB.
5. Random 3D IDB do not detect more prostate cancer than TRUS random biopsies.
6. The rate of re-biopsies is equal between the two groups.
7. There is no correlation of the cytological and histological results.

ELIGIBILITY:
Inclusion criteria

* Patients without previous biopsies.
* Men aged < 75 years, in whom it is clinically relevant to decide whether he has prostate cancer.
* PSA > 3 - 4 ng/ml and < 20 ng/ml.
* Suspicious findings on DRE or TRUS.
* Informed consent.

Exclusion criteria

* Patients who refuse to sign the consent form for any reason or do not accept the study premises.
* Patients who want to withdraw for any reason during the study.
* Patients with contraindications to MRI (pacemaker, claustrophobia etc.)
* Patients who have already undergone a high quality MRI examination of the prostate within the last year. In this situation the MRI examination will be evaluated together with the surgeon and radiologist on an individual basis. In case of a low quality examination, we will disregard the findings, and include the patient.

An accurate record will be kept of all the excluded patients.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cancer detection rate in the two groups | Day 1
  1. Gold standard TRUS biopsies (random biopsies, targeted and overall)
  2. MRI and TRUS fusioned biopsies (random, targeted and overall)

SECONDARY OUTCOMES:
Detection rate of Gleason grade 4 and 5 tumors in the two groups | Day 1
  Positive biopsies will be classified according to Gleason score.
Total length of biopsies and cancer involvement for targeted, random and all biopsies in both groups | day 1
  The length and cancer involvement will be measured of each biopsy
Patient experience of pain during the biopsy and subjective patients perceptions of durations of the biopsy procedure | day 1
  All patients will answer a questionnaire after the procedure.
Difference in biopsy yield for Urologist 1 and Urologist 2 performing the gold standard biopsies | day 1
  As two different urologists are performing all gold standard biopsies, the results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rud, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Aker, Oslo, Norway